CLINICAL TRIAL: NCT00002759
Title: A PHASE I STUDY OF IRINOTECAN (CPT-11) WITH PHARMACOKINETIC MODULATION BY CYCLOSPORINE A AND PHENOBARBITAL
Brief Title: Irinotecan Plus Cyclosporine and Phenobarbital in Treating Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02242; UCCRC-8033; NCI-T95-0100H; CDR0000064707 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-03-26 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2006-05

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Lymphoma; Neutropenia; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; drug/agent toxicity by tissue/organ; neutropenia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Lymphoma; Neutropenia; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclosporine; Irinotecan; Phenobarbital

ARMS (1):
- Arm I (Experimental): See detailed description.
  Interventions: Drug: cyclosporine; Drug: irinotecan hydrochloride; Drug: phenobarbital

INTERVENTIONS:
Drug: cyclosporine
Drug: irinotecan hydrochloride
Drug: phenobarbital

SUMMARY:
Phase I trial to study the effectiveness of irinotecan plus cyclosporine and phenobarbital in treating patients who have solid tumors or lymphoma that is refractory to standard therapy. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Cyclosporine and phenobarbital may enhance the effectiveness of irinotecan.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of irinotecan (CPT-11) when infused weekly with cyclosporine (CYSP) in patients with solid tumors or lymphoma refractory to standard therapy.

II. Determine whether CYSP modulates the pharmacokinetics and pharmacodynamics of CPT-11 and its active metabolite, SN-38.

III. Determine whether phenobarbital modulates the pharmacokinetics and pharmacodynamics of CPT-11 and SN-38.

OUTLINE: This is a dose escalation study of irinotecan. Patients are stratified according to gender.

Part I: Patients receive cyclosporine IV over 6 hours and irinotecan IV over 90 minutes weekly for 4 weeks. Courses repeat every 6 weeks in the absence of unacceptable toxicity or disease progression. Cohorts of 3-12 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least one third of patients experience dose limiting toxicity (DLT).

Part IIA: If the DLT is diarrhea in part I, then part IIA is opened. Patients receive oral phenobarbital, cyclosporine as in part I, and irinotecan at the MTD from part I. Dose escalation occurs as in part I to determine a new MTD. If the DLT continues to be diarrhea, the study is closed. Part IIB: If the DLT is neutropenia in part I, then part IIB is opened. Patients receive cyclosporine as in part I and escalating doses of irinotecan to determine a new MTD.

Part III: If the DLT is neutropenia in part IIA or any DLT in part IIB, patients receive phenobarbital, cyclosporine, and irinotecan at the MTD determined as in part IIA or part IIB. Dose escalation continues until a new MTD is determined.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Malignant solid tumor or lymphoma refractory to standard therapy or for which no therapy of proven benefit exists
* No leukemia
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: Karnofsky 70-100%
* Life expectancy: At least 3 months
* WBC at least 3,500/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9 g/dL
* Bilirubin no greater than 1.5 mg/dL
* AST/ALT less than twice normal (unless due to disease)
* PT and PTT normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No history of congestive heart failure requiring medical therapy
* No clinically significant or life threatening cardiac arrhythmia
* No history of significant pulmonary disease or lymphangitic lung disease
* No hypersensitivity to cyclosporine or cremophore
* No history of manifest or latent porphyria or hypersensitivity to barbiturates (for parts of study using phenobarbital)
* No history of inflammatory bowel disease requiring therapy
* No chronic diarrhea syndrome or paralytic ileus
* No medical or psychiatric condition that precludes informed consent
* Not pregnant
* Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior biologic therapy
* At least 2 weeks since prior colony stimulating factors
* At least 4 weeks since prior chemotherapy (at least 6 weeks since nitrosoureas or mitomycin)
* No prior bleomycin or irinotecan
* At least 4 weeks since prior radiotherapy to greater than 25% of bone marrow
* Minimum time interval between prior therapy and eligibility shortened by 2 weeks when phenobarbital is administered
* Concurrent use of medications that affect the central nervous or cardiovascular systems (e.g., anticonvulsants, calcium channel blockers, oral contraceptives) must be approved by the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 1996-06; Primary Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J. Ratain, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States